CLINICAL TRIAL: NCT05751343
Title: Atezolizumab Plus Bevacizumab Plus Transarterial Chemoembolization and Hepatic Artery Infusion Chemotherapy for Unresectable Advanced Hepatocellular Carcinoma: a Single-arm Phase 2 Clinical Trial
Brief Title: Atezolizumab and Bevacizumab Plus TACE-HAIC for Unresectable Advanced HCC: a Phase 2 Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-141
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The TACE-HAIC which was performed using 30 mg/m2 of epirubicin mixed with 2-5 mL lipiodol, followed by pure lipiodol. Then, a catheter was placed and fixed in the tumor feeding artery for the FOLFOX-based chemotherapy infusion at the following dosage: 85 mg/m2 of oxaliplatin infusion for 2 hours; leucovorin, 400 mg/m2 infusion for 2 hours; 400 mg/m2 of 5-FU bolus; and 1200mg/m2 of continuous 5-FU infusion for 23 hours, respectively. Repeated TACE-HAIC was performed at intervals of 3-4 weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TACE-HAIC plus atezolizumab-bevacizumab (Experimental): transartery chemoembolization and hepatic artery infusion of FOLFOX, simultaneously followed by intravenous of 1200mg atezolizumab plus bevacizumab (15mg/kg)
  Interventions: Drug: TACE-HACI, plus atezolizumab-bevacizumab

INTERVENTIONS:
Drug: TACE-HACI, plus atezolizumab-bevacizumab — transartery chemoembolization and artery infusion of FOLFOX, simultaneously followed by intravenous atezolizumab plus bevacizumab

SUMMARY:
Atezolizumab and bevacizumab was approve for advanced unresectable hepatocellular carcinoma (aHCC). Whether the additional of transartial chemobolization and hepatic artery infusion chemotherapy will improve the response rate for those patients is still unknown. This phase 2 clinical trial aims to investigate the objective response rate for unresectable advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* (a) patients were diagnozied with unresectable advanced-stage HCC,
* (b) Child-Pugh A or B liver function;
* (d) Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* (e) adequate hematologic blood counts (white blood cell count >3ⅹ109/L, absolute neutrophil count >1.5ⅹ109/L, platelet count >10ⅹ109/L, hemoglobin concentration >85 g/L);

Exclusion Criteria:

* (a) severe underlying cardiac, pulmonary, or renal diseases;
* (b) history of a second primary malignant tumor;
* (c) contraindication to either atezolizumab and bevacizumab.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 months
  objective response rate based on RECIST 1.1

SECONDARY OUTCOMES:
objective response rate based mRECIST | 12 months
  objective response rate based on modified RECIST criteria
progress-free survival | 12 months
  Progress-free survival (PFS) was defined from the date of treatment to the first image-confirmed progress based on RECIST 1.1, last follow-up or died.
overall survival | 12 months
  Overall survival was defined from the date of treatment to the date of died or last follow-up
adverse event | 12 months
  adverse event was assessed according to the NCI-CTCAEV 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No